CLINICAL TRIAL: NCT05596838
Title: Long-term Result of Placing Intracorneal Rings in Keratoconus Using Laser
Acronym: STAK
Status: Active, not recruiting | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: STAK
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Intracorneal Ring; Keratoconus; Laser
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient operated at Somain institute with the placement of intracorneal rings: patient operated in the last 10 years on one or both eyes
  Interventions: Procedure: Intracorneal rings placement

INTERVENTIONS:
Procedure: Intracorneal rings placement — Intracorneal rings placement in keratoconus using laser

SUMMARY:
Intracorneal rings are indicated in patients whose central cornea does not present opacity and whose visual acuity is not satisfied despite correction with lenses or linked to an intolerance to lenses.

Surgeries such as crosslinking and intracorneal rings placement are alternatives to corneal transplantation with the expected effects: stabilization of the disease for corneal collagen crosslinking and visual rehabilitation by the placement of intracorneal rings.

The main objective of this study is to evaluate visual benefit1 year after placement of intracorneal rings using laser in keratoconus

ELIGIBILITY:
Inclusion Criteria:

* Patient having received the information notice/non-objection
* Adult man or woman (over 18)
* Failure of a lens fitting adaptation
* Patient with a diagnosis of keratoconus
* Patient operated at Somain institute with the placement of intra-corneal rings

Exclusion Criteria:

* Minor
* Post-lasik ectasia
* Iatrogenic Keratoconus
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient operated at Somain institue with the placement f intra-corneal rings using laser
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) evolution. Visual acuity will be expressed in logMAR. | 1 year
  Evolution of the best corrected visual acuity (BCVA) 1 year after the installation of intra-corneal rings compared to the preoperative value. Visual acuity will be expressed in logMAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Ophtalmique de Somain, Somain, France